CLINICAL TRIAL: NCT06527417
Title: The Effect of Electromyography Triggered Electrical Stimulation on Trunk Balance and Muscle Thickness of Multifidus and Erector Spinae Muscles in Patients With Complete Spinal Cord Injury - A Randomised Controlled Study
Brief Title: Electromyography-Triggered Electrical Stimulation on Trunk Balance and Muscle Thickness in SCI Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Handan Elif Nur BAYRAKTAR, Principal Investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AnkaraCHBilkent-PMR-DRHENY-02
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Spinal Cord Injury Thoracic
Keywords: spinal cord injury; trunk balance; electrical stimulation; multifidus; erector spinae
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Intervention Model Description: In this randomized controlled and prospective study, investigators included 15 participants with complete thoracic spinal cord injury. Investigators divided the participants into two groups, where one group received the electromyography-triggered electrical stimulation applied to the erector spinae and multifidus muscles, and the control group received trunk eccentric exercises only, applied three times a week for four weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electromyography-triggered electrical stimulation (Experimental): EMG ES was applied to the bilateral multifidus and erector spina muscles of the experimental group 3 times a week for 10 minutes in each session for 4 weeks. At the beginning of each session, the participants were instructed to position themselves in a comfortable sitting position.
  EMG ES was performed using six self-adhesive electrodes (37 × 64 mm) and two Neuro Trac Myo Plus Pro devices.
  Interventions: Device: Neuro Trac Myo Plus Pro
- trunk eccentric exercises (Active Comparator): The control group performed back eccentric exercises for 4 weeks, 3 times a week, 3 times in each session.
  Interventions: Other: Trunk eccentric exercises

INTERVENTIONS:
Device: Neuro Trac Myo Plus Pro — Electrical stimulation parameters; stimuli were monophasic, rectangular, stimulus duration 300 µs, frequency 25 Hertz, amplitude was increased up to a maximum of 100 milliampere until contraction was seen.
  Arms: electromyography-triggered electrical stimulation
Other: Trunk eccentric exercises — The control group performed back eccentric exercises for 4 weeks, 3 times a week, 3 times in each session
  Arms: trunk eccentric exercises

SUMMARY:
The aim of this study was to investigate the effect of electromyography (EMG) triggered electrical stimulation (ES) applied to multifidus and erector spinae muscles on trunk balance in patients with complete thoracic spinal cord injury (SCI).

The fundamental questions that investigators want to answer are as follows:

* [question 1]: "Does multifidus and erector spinae EMG ES improve trunk balance in patients with complete SCI?"
* [question 2]: "Does multifidus and erector spinae EMG ES improve muscle thickness in patients with complete SCI?"

DETAILED DESCRIPTION:
Spinal cord injury results in loss of sensory and motor function below the level of injury, causing difficulty with unaided sitting and activities of daily living, especially at the thoracic level in SCI patients. The paraspinal muscles that provide trunk balance are weakened in these patients. Methods such as neuromuscular electrical stimulation and EMG ES are used to improve trunk balance and restore muscle function. This study aims to investigate the effect of EMG ES applied to the multifidus and erector spinae muscles on trunk balance in patients with complete thoracic SCI.

ELIGIBILITY:
Inclusion Criteria:

* have traumatic SCI and this injury occurred at least 3 months ago,
* be between the ages of 18 and 65,
* have a neurological injury level between thoracic 4 and thoracic 12
* be fully paraplegic according to the American Spinal Cord Injury Association (ASIA) impairment scale
* be able to sit unsupported in a wheelchair

Exclusion Criteria:

* patients with a diagnosis of heart failure
* malignancy
* intracardiac defibrillators
* epilepsy
* open wounds
* patients using trunk corsets

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-08-18 (Actual); Primary Completion 2024-02-18 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Trunk control test | Baseline- Week 4
  The trunk control test is a useful tool in determining the prognosis of independence in activities of daily living and measuring trunk balance in individuals with spinal cord injury. It was applied to all participants before and after treatment. The test consisted of 3 parts; static control, dynamic control and dynamic control with upper extremity activities.
Modified functional reach test | Baseline- Week 4
  The modified functional reach test is a reliable tool to assess sitting reaching in individuals with SCI and to provide immediate feedback to study personnel. It was applied to both groups before and after treatment.

SECONDARY OUTCOMES:
Erector spinae muscle thickness | Baseline- Week 4
  Erector spinae muscle thickness was measured with a real-time B-mode ultrasound device (General Electric Co., Wisconsin, USA). Measurements were performed bilaterally in the prone position with an 8-12 MegaHertz linear probe placed parallel to the muscle fibres. Gel was used between the probe and the skin during the measurements. The measurement site was defined as 7 cm lateral to the L3 spinous process of the lumbar erector spina muscle.

OTHER OUTCOMES:
Multifidus muscle thickness | Baseline- Week 4
  Multifidus muscle thickness was measured with a real-time B-mode ultrasound device (GE, General Electric Co., Wisconsin, USA). Measurements were performed bilaterally in the prone position with an 8-12 MegaHertz linear probe placed parallel to the muscle fibres. Gel was used between the probe and the skin during the measurements. The measurement site was defined as 2 cm lateral to the L4 spinous process of the Multifidus muscle.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bjerkefors A, Carpenter MG, Cresswell AG, Thorstensson A. Trunk muscle activation in a person with clinically complete thoracic spinal cord injury. J Rehabil Med. 2009 Apr;41(5):390-2. doi: 10.2340/16501977-0336. PMID 19363574
- [Background] Bergmann M, Zahharova A, Reinvee M, Asser T, Gapeyeva H, Vahtrik D. The Effect of Functional Electrical Stimulation and Therapeutic Exercises on Trunk Muscle Tone and Dynamic Sitting Balance in Persons with Chronic Spinal Cord Injury: A Crossover Trial. Medicina (Kaunas). 2019 Sep 21;55(10):619. doi: 10.3390/medicina55100619. PMID 31546613
- [Background] Gill M, Linde M, Fautsch K, Hale R, Lopez C, Veith D, Calvert J, Beck L, Garlanger K, Edgerton R, Sayenko D, Lavrov I, Thoreson A, Grahn P, Zhao K. Epidural Electrical Stimulation of the Lumbosacral Spinal Cord Improves Trunk Stability During Seated Reaching in Two Humans With Severe Thoracic Spinal Cord Injury. Front Syst Neurosci. 2020 Nov 19;14:79. doi: 10.3389/fnsys.2020.569337. eCollection 2020. PMID 33328910
- [Background] Shima D, Nishimura Y, Hashizaki T, Minoshima Y, Yoshikawa T, Umemoto Y, Kinoshita T, Kouda K, Tajima F, Kamijo YI. Surface electromyographic activity of the erector spinae and multifidus during arm- and leg-ergometer exercises in young healthy men. Front Physiol. 2022 Nov 25;13:974632. doi: 10.3389/fphys.2022.974632. eCollection 2022. PMID 36505070
- [Background] Wilson RD, Page SJ, Delahanty M, Knutson JS, Gunzler DD, Sheffler LR, Chae J. Upper-Limb Recovery After Stroke: A Randomized Controlled Trial Comparing EMG-Triggered, Cyclic, and Sensory Electrical Stimulation. Neurorehabil Neural Repair. 2016 Nov;30(10):978-987. doi: 10.1177/1545968316650278. Epub 2016 May 24. PMID 27225977
- [Background] Triolo RJ, Bailey SN, Foglyano KM, Kobetic R, Lombardo LM, Miller ME, Pinault G. Long-Term Performance and User Satisfaction With Implanted Neuroprostheses for Upright Mobility After Paraplegia: 2- to 14-Year Follow-Up. Arch Phys Med Rehabil. 2018 Feb;99(2):289-298. doi: 10.1016/j.apmr.2017.08.470. Epub 2017 Sep 9. PMID 28899825
- [Background] Qiu S, Draghici AE, Picard G, Taylor JA. Muscle Fatigue in Response to Electrical Stimulation Pattern and Frequency in Spinal Cord Injury. PM R. 2020 Jul;12(7):699-705. doi: 10.1002/pmrj.12282. Epub 2019 Dec 12. PMID 31702873
- [Background] Tharu NS, Alam M, Ling YT, Wong AY, Zheng YP. Combined Transcutaneous Electrical Spinal Cord Stimulation and Task-Specific Rehabilitation Improves Trunk and Sitting Functions in People with Chronic Tetraplegia. Biomedicines. 2022 Dec 23;11(1):34. doi: 10.3390/biomedicines11010034. PMID 36672542
- [Background] Lee HS, Akimoto T, Kim AR. Effects of trunk extensor eccentric exercise on lipid profile and glycaemic response. BMJ Open Sport Exerc Med. 2020 Oct 28;6(1):e000861. doi: 10.1136/bmjsem-2020-000861. eCollection 2020. PMID 33178444
- [Background] Quinzanos-Fresnedo J, Fratini-Escobar PC, Almaguer-Benavides KM, Aguirre-Guemez AV, Barrera-Ortiz A, Perez-Zavala R, Villa-Romero AR. Prognostic validity of a clinical trunk control test for independence and walking in individuals with spinal cord injury. J Spinal Cord Med. 2020 May;43(3):331-338. doi: 10.1080/10790268.2018.1518124. Epub 2018 Sep 12. PMID 30207875
- [Background] Arsh A, Darain H, Rahman MU, Ullah I, Shakil-Ur-Rehman S. Reliability of modified functional reach test in the assessment of balance function in people with spinal cord injury: A systematic review. J Pak Med Assoc. 2021 Aug;71(8):2040-2044. doi: 10.47391/JPMA.1276. PMID 34418026
- [Background] Masaki M, Aoyama T, Murakami T, Yanase K, Ji X, Tateuchi H, Ichihashi N. Association of low back pain with muscle stiffness and muscle mass of the lumbar back muscles, and sagittal spinal alignment in young and middle-aged medical workers. Clin Biomech (Bristol). 2017 Nov;49:128-133. doi: 10.1016/j.clinbiomech.2017.09.008. Epub 2017 Sep 14. PMID 28934633
- [Background] Masaki M, Ikezoe T, Fukumoto Y, Minami S, Tsukagoshi R, Sakuma K, Ibuki S, Yamada Y, Kimura M, Ichihashi N. Association of sagittal spinal alignment with thickness and echo intensity of lumbar back muscles in middle-aged and elderly women. Arch Gerontol Geriatr. 2015 Sep-Oct;61(2):197-201. doi: 10.1016/j.archger.2015.05.010. Epub 2015 May 28. PMID 26058723
- [Background] Bayraktar HEN, Yalcin E, Sipal MS, Akyuz M, Akinci MG, U Delialioglu S. The effect of electromyography triggered electrical stimulation to abdominal muscles on sitting balance, respiratory functions, and abdominal muscle thickness in complete spinal cord injury: a randomized controlled trial. Int J Rehabil Res. 2024 Jun 1;47(2):87-96. doi: 10.1097/MRR.0000000000000620. Epub 2024 Mar 19. PMID 38501227